CLINICAL TRIAL: NCT06686537
Title: Convergent Mechanisms Underlying Reprometabolic Syndrome in Women and Sheep
Brief Title: Convergent Mechanisms Underlying Reprometabolic Syndrome in Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-1269; CO-C-24-218 (Other: U of Colorado CCTSI)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Infertility, Female; Obesity
Keywords: Obesity; Infertility; Hypothalamic-pituitary-ovarian axis; pituitary dysfunction
MeSH Terms: conditions — Infertility, Female; Obesity; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Estradiol Patch- Normal Weight women (Experimental): Normal weight women (NWW) will wear a Transdermal estradiol patch for 7 days and collect urine to determine LH surge.
  Interventions: Drug: Estradiol Patches
- Estradiol Patch- Women with high BMI (Experimental): Women with a BMI greater than 30 kg/m2 will wear a Transdermal estradiol patch for 7 days and collect urine to determine LH surge.
  Interventions: Drug: Estradiol Patches

INTERVENTIONS:
Drug: Estradiol Patches — Estradiol patched will be worn for 7 days.

SUMMARY:
Dr. Nanette Santoro proposes to test the specific question that obesity results in abnormal estradiol response at the level of the pituitary and hypothalamus. This will be shown in diminished pituitary sensitivity to gonadorelin releasing hormone with a reduced estradiol induced luteinizing hormone surge in obese women.

DETAILED DESCRIPTION:
This is an open-label, single site study in pre-menopausal women aged 18-40 years old with a history of regular menstrual cycles (25-35 days long) of normal BMI or high BMI. The objective of the study is to determine the effects of an estradiol patch on luteinizing hormone rise in both cohorts. The study consists of 2 periods: a screening period of up to 3 weeks and a Treatment Period of 7-10 days. During the treatment period participants will wear estradiol patches for up to 7 days and have on blood draw on day 3 of wearing the patches. Participants will also collect daily morning urine for all the days they wear the patches. Participants will use a reliable barrier method of birth control or abstain from intercourse for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-38
* Regular menstrual cycles every 25-35 days
* No use of reproductive hormones within the past 3 months
* No use of medications interacting with reproductive hormones
* Agreement to use reliable barrier contraception or to abstain from intercourse for the duration of the study
* Normal thyroid stimulating hormone, prolactin and lipid profiles
* No more than 4 hours of moderate to vigorous intensity exercise per week
* No history of chronic disease impacting reproductive hormones
* No contraindications to administration of estradiol
* No history of estrogen dependent cancer
* Negative pregnancy test

Exclusion Criteria:

* Has diabetes
* Is a smoker
* History of venous thromboembolism or known thrombophilia

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is limited to only female (assigned at birth) participants due to the requirement for menstruating females.
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Amount of Luteinizing hormone Surge | From enrollment to the end of treatment is 7 days.
  Urinary luteinizing hormone concentration in mIU/mg of Creatinine

SECONDARY OUTCOMES:
Time of Luteinizing Hormone Peak | From enrollment to 7 days
  Specific day of highest urinary luteinizing hormone concentration (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado School of Medicine
Locations (2):
- United States (2):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Colorado-School of Medicine, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain A, Polotsky AJ, Rochester D, Berga SL, Loucks T, Zeitlian G, Gibbs K, Polotsky HN, Feng S, Isaac B, Santoro N. Pulsatile luteinizing hormone amplitude and progesterone metabolite excretion are reduced in obese women. J Clin Endocrinol Metab. 2007 Jul;92(7):2468-73. doi: 10.1210/jc.2006-2274. Epub 2007 Apr 17. PMID 17440019
- [Background] Rovner P, Keltz J, Allshouse A, Isaac B, Hickmon C, Lesh J, Chosich J, Santoro N. Induction of the LH Surge in Premenarchal Girls Confirms Early Maturation of the Hypothalamic-Pituitary-Ovarian Axis. Reprod Sci. 2018 Jan;25(1):33-38. doi: 10.1177/1933719117741377. Epub 2017 Nov 19. PMID 29153058